CLINICAL TRIAL: NCT06973057
Title: Direct Pulp Capping Versus Pulpotomy Using Neo MTA for Carious Primary Molars: a Split Mouth Randomized Clinical Trial
Brief Title: Direct Pulp Capping Versus Pulpotomy for Primary Molars
Acronym: MTA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 341-2023
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Vital Pulp Therapies
Keywords: Vital Pulp therapies; Direct pulp capping; Pulpotomy; Neo MTA; Primary molars; Randomized clinical trial
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: A split mouth randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Active Comparator): The entire coronal pulp will be amputated.
  Interventions: Procedure: Pulpotomy
- Direct pulp capping (Active Comparator): The exposure site will be left intact, no amputation of pulp tissue.
  Interventions: Procedure: Direct pulp capping (DPC)

INTERVENTIONS:
Procedure: Pulpotomy — The entire coronal pulp will be amputated to the level of canal orifices, after hemostasis, NeoMTA will be placed, then tooth will be restored with glass ionomer cement, and the tooth will be subsequently restored with a crown.
  Arms: Pulpotomy
Procedure: Direct pulp capping (DPC) — At the exposure site hemostasis will be achieved, neo MTA will be placed, then tooth will be restored with glass ionomer cement, and the tooth will be subsequently restored with a crown.
  Arms: Direct pulp capping

SUMMARY:
Dental caries is one of the most prevalent chronic diseases worldwide. Interventions for treating deep carious lesions in teeth with no history of pain or teeth with reversible pulpitis are referred to as vital pulp therapy; these include indirect pulp treatment (IPC), direct pulp capping (DPC), and pulpotomy. Pulpotomy is considered invasive when treating exposed primary vital pulps due to caries. Less invasive vital pulp treatment methods such as DPC might, therefore, be preferable, as they reduce chair time, less tooth structure removal and a crown might not always be a necessary permanent restoration. The aim of this clinical study is to evaluate the clinical and radiographic outcomes of DPC when compared to pulpotomy in primary molars with carious pulp exposure.

DETAILED DESCRIPTION:
Aim: The aim of this study is to evaluate the clinical and radiographic outcomes of direct pulp capping (DPC) when compared to pulpotomy in primary molars with carious pulp exposure using a calcium silicate-based material: neo mineral trioxide aggregate (Neo MTA).

Methods: The study will be a split mouth randomized clinical trial including children between 4-9 years old. Patients will be allocated into two treatment groups; one group will start with DPC first followed by pulpotomy on the second visit, and vice versa for the second group. The time interval between both visits will be 1-2 weeks. The pulp medicament capping material (neo MTA) will be applied over the exposure site, and then tooth will be restored with glass ionomer cement and then a crown will be placed. Cases will be followed up to 24 months after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients.
* Age 4-10 years.
* Primary molar with deep caries present bilaterally.
* Teeth should be restorable.
* Clinically normal asymptomatic tooth or symptoms of reversible pulpitis (No history of pain or provoked pain subsides upon removal of the stimulus).
* Radiographically: caries in the inner half of the dentin approaching the pulp.

Exclusion Criteria:

* History of spontaneous pain.
* Soft and hard tissue pathology.
* Mobility or exfoliating tooth.
* No pulp exposure after caries excavation.
* Inability to achieve hemostasis after 6 minutes.
* Radiographically: Root resorption exceeding 1/3 of the root, apical pathology.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 24 months
  No post-treatment signs or symptoms such as sensitivity, pain, mobility or swelling should be evident.
Radiographic success | 24 months
  No radiographic evidence of pathologic external or internal root resorption, periapical or furcation radiolucency.

CONTACTS AND LOCATIONS:
Overall Officials: OLA Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan Univeristy of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dimitraki D, Papageorgiou SN, Kotsanos N. Direct pulp capping versus pulpotomy with MTA for carious primary molars: a randomised clinical trial. Eur Arch Paediatr Dent. 2019 Oct;20(5):431-440. doi: 10.1007/s40368-019-00419-7. Epub 2019 Feb 20. PMID 30788777
- [Result] Alsanouni M, Bawazir OA. A Randomized Clinical Trial of NeoMTA Plus in Primary Molar Pulpotomies. Pediatr Dent. 2019 Mar 15;41(2):107-111. PMID 30992107
- [Result] ElSebaai A, Wahba AH, Grawish ME, Elkalla IH. Calcium Hydroxide Paste, Mineral Trioxide Aggregate, and Formocresol as Direct Pulp Capping Agents in Primary Molars: A Randomized Controlled Clinical Trial. Pediatr Dent. 2022 Nov 15;44(6):411-417. PMID 36947754
- [Result] Chatzidimitriou K, Vadiakas G, Koletsi D. Direct pulp capping in asymptomatic carious primary molars using three different pulp capping materials: a prospective clinical trial. Eur Arch Paediatr Dent. 2022 Oct;23(5):803-811. doi: 10.1007/s40368-022-00720-y. Epub 2022 Jul 2. PMID 35780237
- [Result] Canoglu E, Gungor HC, Uysal S. Direct Pulp Capping of Primary Molars with Calcium Hydroxide or MTA Following Hemorrhage Control with Different Medicaments: Randomized Clinical Trial. Pediatr Dent. 2022 May 15;44(3):167-173. PMID 35799339
- See also: Pulp Therapy for Primary and Immature Permanent Teeth — https://www.aapd.org/media/Policies_Guidelines/BP_PulpTherapy.pdf